CLINICAL TRIAL: NCT04802122
Title: Comparative Assessment of Intubating Conditions and Cardiorespiratory Effects of Sevoflurane Induction and Intubation.
Brief Title: Induction of Anesthesia With Sevoflurane Preserving Spontaneous Breathing: Cardiorespiratory Effects.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Georgia Tsaousi, Associate Professor, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INTUSEVO
Record Dates: First submitted 2021-03-14; First posted 2021-03-17 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Anesthesia Intubation Complication; Cardiovascular Complication; Intubation
Keywords: inhalational; sevoflurane; cardiovascular; induction
MeSH Terms: interventions — Sevoflurane; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sevoflurane group (Experimental): Patients in this group will receive Sevoflurane 8% / O2 100% with the vital capacity breathing method (vital capacity induction, VCI) for induction to anesthesia and to facilitate endotracheal intubation (without the use of muscle relaxant) and thereafter Sevoflurane 1 MAC will be used for maintenance of anesthesia plus muscle relaxant until study completion.
  Interventions: Drug: Sevoflurane inhalant product
- Propofol group (Active Comparator): Patients in this group will receive a standard anesthesia induction involving Propofol 1,5mg/Kg, supplemented by fentanyl 2mcg/Kg and rocuronium 0,5mg/Kg and O2 100% for induction to anesthesia and to facilitate endotracheal intubation and thereafter Sevoflurane 1 MAC will be used for maintenance of anesthesia.
  Interventions: Drug: Propofol Fresenius

INTERVENTIONS:
Drug: Sevoflurane inhalant product — Sevoflurane 8% / O2 100% with the vital capacity breathing method (vital capacity induction, VCI) will be used for induction to anesthesia and facilitate endotracheal intubation.
  Other Names: Sevoflurane
  Arms: Sevoflurane group
Drug: Propofol Fresenius — Propofol 1,5mg/Kg, supplemented by fentanyl 2mcg/Kg and rocuronium 0,5mg/Kg and O2 100% will be for induction to anesthesia and facilitate endotracheal intubation. .
  Other Names: Propofol
  Arms: Propofol group

SUMMARY:
Airway management is of outmost importance in the perioperative period. One of the main questions while making a plan for airway management is whether spontaneous ventilation should be maintained or not. Induction of anesthesia with Sevoflurane is a conventional technique that preserves spontaneous ventilation. It is used especially in non-collaborating patients or when other pharmaceutical agents or sophisticated airway management equipment is out of reach.

Inhalational induction of anesthesia with Sevoflurane is well studied. However, there are few studies investigating the effects of Sevoflurane on induction and intubating conditions, on cardiopulmonary physiology, on emergence conditions, when it is used as one and only agent to achieve induction of anesthesia, intubation and maintenance of anesthesia in adult patients. There is also no consensus on the appropriate duration of the inhalational induction or other criteria to guarantee successful intubation conditions, since most studies investigate Sevoflurane administration until induction of anesthesia and not until intubation.

From all the above, it appears that there are a few gaps in the management of patients who are to be intubated with Sevoflurane only, without the use of any other anesthetic agents.

DETAILED DESCRIPTION:
Preoperatively, the study protocol-mandated baseline data will be recorded: gender, age, body weight, body mass index, body surface area, ASA-PS, type of surgery. The airway assessment will include Mallampati score, thyromental distance, cervical spine mobility, upper lip bite test, mouth opening, micrognathia, protruding incisors, beard, denture, snoring.

Patients will be randomly allocated into one of two groups: the S group was to be intubated after inhalational anesthesia with Sevoflurane only and maintenance of anesthesia with Sevoflurane 1MAC. The P group will receive standard anesthesia induction with propofol 1,5mg/Kg, fentanyl 2mcg/Kg, rocuronium 0,5mg/Kg, while anesthesia will be maintained by sevoflurane.

Before induction of anesthesia, we will record baseline data including BIS, SpO2, heart rate, invasive blood pressure, cardiac output, stroke volume, stroke volume variation, respiratory rate, and arterial blood gas sample recordings.

During induction of anesthesia, the following data will be recorded: BIS, SpO2, heart rate, invasive blood pressure, cardiac output, stroke volume, stroke volume variation, respiratory rate, recordings from arterial blood gas sample, induction to anesthesia conditions (limb movement, cough, salivation, laryngospasm, and apnea), respiratory rate, tidal volume, minute volume, end-tidal CO2, the concentration of sevoflurane (inhaled, exhaled), peak inspiratory pressure, mean inspiratory pressure, dynamic respiratory compliance. In the S group, these data will be recorded again five minutes after the induction to anesthesia commencement.

During intubation, we will record BIS, SpO2, heart rate, blood pressure, cardiac output, stroke volume, stroke volume variation, intubating conditions (jaw relaxation, vocal cord position, vocal cord movement, limb movement, bucking), Cormack-Lehane grade, duration of intubation.

After intubation we will register: BIS, SpO2, heart rate, invasive blood pressure, cardiac output, stroke volume, stroke volume variation, respiratory rate, recordings from arterial blood gas sample, respiratory rate, tidal volume, minute volume, end-tidal CO2, the concentration of sevoflurane (inhaled, exhaled), peak inspiratory pressure, mean inspiratory pressure, dynamic respiratory compliance, were recorded. Patients having abolished spontaneous breathing will be set on the IMV mode of ventilation receiving tidal volume 8ml/Kg, 10 breaths/min, PEEP=5cmH2O, I: E=1:2, Plateau time 30%.

Upon the end of the surgical stimuli the following parameters will be registered: BIS, blood pressure, heart rate, SpO2, stroke volume, stroke volume variation, cardiac output, etCO2, respiratory rate, sevoflurane concentration (exhaled, inhaled), peak inspiratory pressure, mean inspiratory pressure, dynamic compliance, time of establishing spontaneous breathing, time of extubation.

BIS, blood pressure, heart rate, SpO2, stroke volume, stroke volume variation, cardiac output, etCO2, the respiratory rate will be recorded 5 and 10 minutes respectively post-extubation.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 and < 71 years
* ASA-PS 1-3 (American Society of Anesthesiologists Physical Status classification)
* General anesthesia for abdominal surgery
* Elective cases
* Signed informed consent

Exclusion Criteria:

* Urgent/emergency surgeries
* BMI<18.5 or BMI>34.9
* Intraabdominal hypertension
* Gastroesophageal reflex
* Pregnancy
* Liver or renal failure
* intracranial hypertension

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-05-24 (Actual); Primary Completion 2021-07-13 (Actual); Study Completion 2021-07-14 (Actual)

PRIMARY OUTCOMES:
Intubating conditions | 10 minutes after induction to anesthesia commencement with sevoflurane or 5 minutes after induction to anesthesia with propofol plus fentanyl and muscle relaxant
  Modification of intubating conditions assessed by Cormack-Lehane classification system after induction to anesthesia with sevoflurane (without muscle relaxants) or standard induction to anesthesia involving propofol supplemented by fentanyl and muscle relaxant.
Cardiac output compromise | Within 10 minutes after induction to anesthesia commencement with sevoflurane or 5 minutes after induction to anesthesia with propofol plus fentanyl and muscle relaxant
  Cardiac index reduction defined CI < 2.2 L/min/m2 after induction to anesthesia with sevoflurane (without muscle relaxants) or standard induction to anesthesia involving propofol supplemented by fentanyl and muscle relaxant.

SECONDARY OUTCOMES:
Hypercapnia | 1 minute after intubation
  The occurrence of hypercapnia defined as carbon dioxide partial pressure > 45 mmHg in arterial blood gas sample after induction to anesthesia with sevoflurane (without muscle relaxants) or standard induction to anesthesia involving propofol supplemented by fentanyl and muscle relaxant.
Hypotension | Within10 minutes after induction to anesthesia commencement with sevoflurane or 5 minutes after induction to anesthesia with propofol plus fentanyl and muscle relaxant
  Duration of hypotension defined as systemic arterial pressure < 90mmHg after induction to anesthesia with sevoflurane (without muscle relaxants) or standard induction to anesthesia involving propofol supplemented by fentanyl and muscle relaxant.

CONTACTS AND LOCATIONS:
Overall Officials: Vasilios Grosomanidis, Study Director — Aristotle University Of Thessaloniki
Locations (1):
- AHEPA University Hospital, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No